CLINICAL TRIAL: NCT06832592
Title: Etude Descriptive Des Besoins en Soins de Support Des Patients en Phase Active de Traitement d'un Cancer Bronchique en Oncologie Ambulatoire à l'hôpital Nord-Ouest de Villefranche/Saône.
Brief Title: Supportive Care Needs of Bronchial Cancer Patients in Active Treatment: A Descriptive Study in Outpatient Oncology
Status: Completed | Type: Observational
Sponsor: L'hôpital Nord-Ouest - Villefranche Villefranche sur Saône (Other)
Responsible Party: Sponsor
Other Study IDs: HNO24_001
Record Dates: First submitted 2025-02-07; First posted 2025-02-18 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-02

CONDITIONS: Lung Carcinoma
Keywords: Lung cancer; Supportive oncological care; Patient needs; Self-questionnaire
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- SOS-LUNG: population of 100 adults followed in the outpatient oncology department for lung cancer who are given a self-questionnaire on their need for supportive care after delivery of an information notice and collection of their non-opposition, over the period from February to April 2025.

SUMMARY:
Bronchial cancer is a major oncological pathology, representing the leading cause of cancer death in France. Supportive oncological care (SOS) is defined as all the care and support necessary for patients throughout their journey, in addition to specific treatments. Despite their importance, their identification and accessibility remain heterogeneous in outpatient oncology. This single-center observational study aims to describe the supportive care needs of patients with bronchial cancer in the active phase of treatment at the Nord-Ouest Hospital in Villefranche-sur-Saône. A self-questionnaire based on the national SOS identification grid will be offered to 100 patients followed in thoracic oncology. The main objective is to identify priority needs perceived and expressed by patients, particularly in terms of psychological support, pain management, nutrition, physical activity, fatigue and social impact. Secondary objectives include the evaluation of the proposal and acceptance of SOS by patients, the analysis of the causes of refusal and the study of variations in needs according to the temporality of treatments and demographic characteristics. A descriptive statistical analysis will be carried out, supplemented by comparative tests to explore the relationships between identified needs and patient profiles. The expected results will make it possible to optimize the provision of supportive care in outpatient oncology, by proposing strategies adapted to the specific needs of patients with bronchial cancer.

DETAILED DESCRIPTION:
Bronchial cancer is a leading oncological pathology, representing the leading cause of cancer death in France. In 2023, there were 52,777 new cases, with a downward trend in men but a notable increase in women. Despite therapeutic advances, this pathology remains associated with high morbidity and a significant impairment of patients' quality of life. Supportive oncological care is defined as all the care and support necessary for patients throughout their journey, in addition to specific oncological treatments. The national framework for supportive oncological care (2021) highlights their essential role in improving the quality of life of patients with cancer, but their evaluation and proposal remain heterogeneous, particularly in outpatient oncology. In this context, this single-center observational study aims to describe the supportive care needs of patients with bronchial cancer in the active phase of treatment at the Nord-Ouest Hospital in Villefranche-sur-Saône.

A self-questionnaire inspired by the national grid for identifying supportive oncological care will be offered to 100 patients followed in thoracic oncology. The main objective is to identify priority supportive care needs, whether perceived by professionals or expressed directly by patients. This identification will concern several areas: understanding the disease and treatments, pain management, psychological support, nutrition, physical activity, fatigue, sleep, maintaining social and professional life, sexuality and lifestyle habits. The study will also focus on the supportive care actually offered and its acceptance by patients, in order to assess possible disparities between the needs identified and the existing offer.

Secondary objectives include the analysis of the causes of refusal of supportive care, the evaluation of patient satisfaction with the existing offer and the study of the influence of the temporality of treatments on the evolution of needs. The study will also seek to determine whether these needs vary based on certain demographic characteristics such as age and gender.

From a methodological point of view, the data will be analyzed using a descriptive and comparative approach. The results will be expressed in frequencies and percentages for qualitative variables, and in means or medians for quantitative variables. Appropriate statistical tests will make it possible to compare groups and identify factors influencing the variability of needs.

The study will take place over a period of one month, with inclusion planned for February 2025 and completion in March 2025. Each patient will participate in the study over a single day, corresponding to the completion of the self-questionnaire during an outpatient oncology consultation. The questionnaire will be distributed by the investigator and can be completed with the help of a caregiver if necessary.

The expected results will make it possible to optimize the provision of outpatient oncology supportive care, by identifying unmet needs and obstacles to access to this care. They could also contribute to the implementation of improvement strategies adapted to the specificities of patients with bronchial cancer, in order to ensure more complete and personalized care.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with bronchial cancer in the active phase of treatment followed in the Ambulatory Oncology department of HNO Villefranche sur Saône.
2. Major
3. Knowing how to read and write French
4. Affiliate to a Social Security scheme

Exclusion Criteria:

1. Patient with cognitive disorder(s)
2. Person under guardianship, curatorship or legal protection
3. Patient objecting to participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient suffering from lung cancer and followed in the outpatient oncology department of the HNOV
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
Proportion of Patients Reporting Unmet Supportive Care Needs Using a Standardized Identification Grid. | At the time of outpatient consultation (Day 0)
  Assessment of supportive care needs in patients with bronchial cancer using a standardized first-level identification grid. Needs will be categorized (e.g., psychological, nutritional, pain management, social support) and reported as the proportion of patients identifying at least one unmet need in each category.

SECONDARY OUTCOMES:
Evaluate whether supportive care is offered by the healthcare team and accepted by patients. | At the time of outpatient consultation (Day 0)
  Binary judgment criteria (yes/no) to additional questions added to the INCA reference grid
Analyze the causes of refusal of help by patients and evaluate the satisfaction of the supportive care offer | At the time of outpatient consultation (Day 0)
  Answers to questions about the benefit of meeting a professional; managing the situation without help; sufficient advice and open responses and the rate of "unsatisfied" patient responses less than 5%

CONTACTS AND LOCATIONS:
Overall Officials: ODIER LUC, Lung Doctor, Study Director — Hôpitaux Nord-Ouest Villefranche Sur Saône
Locations (1):
- HNO Villefranche, Gleizé, France

IPD SHARING:
Plan to Share IPD: Undecided
compliance with the regulations of the Data Protection Act, no transfer to the EU to respect the commitment to conform to the CNIL reference methodology MR-03.